CLINICAL TRIAL: NCT00003972
Title: A Phase III Study of High-Dose Chemotherapy Using Busulfan, Melphalan and Thiotepa Versus Cyclophosphamide,Thiotepa, Carboplatin Followed by Autologous Stem Cell Transplantation in Patients With High-Risk Primary Stage II or III (Non-Inflammatory) Breast Cancer
Brief Title: Combination Chemotherapy and Peripheral Stem Cell Transplantation in Treating Patients With Stage II or Stage IIIA Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 1316.00; FHCRC-1316.00; PSOC-1604; NCI-G99-1552; CDR0000067175 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-05-03 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; sargramostim; Busulfan; Carboplatin; Cyclophosphamide; Melphalan; Paclitaxel; Tamoxifen; Thiotepa; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Biological: sargramostim
Drug: busulfan
Drug: carboplatin
Drug: cyclophosphamide
Drug: melphalan
Drug: paclitaxel
Drug: tamoxifen citrate
Drug: thiotepa
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. It is not yet known which regimen of combination chemotherapy is more effective for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two regimens of combination chemotherapy followed by peripheral stem cell transplantation in treating patients who have stage II or stage IIIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare early mortality, survival, and disease free survival in patients with node positive stage II or IIIA breast cancer treated with busulfan, melphalan, and thiotepa versus cyclophosphamide, thiotepa, and carboplatin followed by autologous peripheral blood stem cell transplantation. II. Compare the toxicity of these 2 regimens in this patient population.

OUTLINE: This is a randomized study. Patients are stratified according to stage of disease (stage II vs stage IIIA), lymph node status (at least 10 positive nodes vs less than 10 positive nodes), and hormone receptor status (estrogen receptor positive or progesterone receptor positive vs estrogen receptor negative or progesterone receptor negative). All patients initially receive mobilization chemotherapy with cyclophosphamide IV over 1-2 hours on day 1 and paclitaxel IV over 4 hours on day 2. Beginning on day 4, patients receive filgrastim (G-CSF) or sargramostim (GM-CSF) subcutaneously each day until the final day of leukapheresis. When blood counts recover, peripheral blood stem cells (PBSC) are harvested. Patients are randomized to 1 of 2 high dose chemotherapy regimens 28-45 days after the last dose of mobilization chemotherapy. Arm I: Patients receive oral busulfan every 6 hours on days -8 to -6, melphalan IV over 30-60 minutes on days -5 and -4, and thiotepa IV over 2 hours on days -3 and -2. PBSC are reinfused on day 0. Arm II: Patients receive cyclophosphamide, thiotepa, and carboplatin by continuous IV infusion over 24 hours on days -7, to -4. PBSC are reinfused on day 0. Beginning 4-6 weeks after the last dose of chemotherapy, patients in both arms receive local radiotherapy 5 days each week for 5 weeks. Patients also receive oral tamoxifen (or equivalent antiestrogen therapy) daily for 5 years if they are estrogen or progesterone receptor positive, postmenopausal, or age 50 and over and perimenopausal. Patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 280 patients (140 per treatment arm) will be accrued for this study over 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage II breast cancer with 1 of the following: Estrogen receptor negative with at least 4 positive nodes OR Estrogen receptor positive with at least 6 positive nodes OR Histologically proven stage IIIA breast cancer Must have already received 4-7 courses of conventional chemotherapy with a doxorubicin based regimen (which may include paclitaxel or docetaxel) No greater than 60 days since induction chemotherapy Prior definitive surgical treatment of primary lesion (modified radical mastectomy or breast conserving procedure plus axillary node dissection) Margins free of tumor Hormone receptor status: Estrogen and progesterone receptor status known

PATIENT CHARACTERISTICS: Age: 18 to 65 Menopausal status: Not specified Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT or SGPT no greater than 2 times normal Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: Left ventricular ejection fraction at least 50% if any of the following: Symptoms of congestive heart failure Abnormal cardiac exam Prior doxorubicin dose greater than 400 mg/m2 Pulmonary: No significant pulmonary disease (DLCO less than 60% predicted) Other: Not pregnant Negative pregnancy test HIV negative No significant active infection No other severe disease that would severely limit life expectancy No other malignancy within past 5 years unless: Chance of survival for greater than 5 years is 90% AND Treated with surgery only (no chemotherapy or radiotherapy)

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No greater than 1 prior chemotherapy regimen (no greater than 7 prior courses) Endocrine therapy: No concurrent tamoxifen Radiotherapy: Not specified Surgery: See Disease Characteristics Other: No other concurrent experimental agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 1998-07; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William I. Bensinger, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States